CLINICAL TRIAL: NCT00399503
Title: Risk Estimation Following Infarction Noninvasive Evaluation (REFINE)
Brief Title: Assessment of Noninvasive Methods to Identify Patients at Risk of Serious Arrhythmias After a Heart Attack
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); Alberta Heritage Foundation for Medical Research (Other); GE Healthcare (Industry); Cambridge Heart Inc. (Industry); Hoffmann-La Roche (Industry)
Other Study IDs: CIHR 73-1518; HSFA 73-1220
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2006-11

CONDITIONS: Myocardial Infarction; Death, Sudden, Cardiac; Death
Keywords: Noninvasive assessment; Combined parameter; Holter
MeSH Terms: conditions — Myocardial Infarction; Death, Sudden, Cardiac; Death

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Spectral T Wave Alternans
Procedure: Modified Moving Average T Wave Alternans
Procedure: Baroreceptor Sensitivity
Procedure: Heart Rate Variability
Procedure: Heart Rate Turbulence
Procedure: Deceleration Capacity
Procedure: Signal Averaged ECG

SUMMARY:
This study evaluates the usefulness of noninvasive tests of the structure of the heart and the nervous system controlling the heart. It will assess whether combining tests that evaluate heart structure with others that measure the nervous system controlling the heart will identify most patients who develop serious heart rhythm problems after a heart attack.

DETAILED DESCRIPTION:
Background. Sudden cardiac death (SCD) kills >450,000 North Americans each year. Patients with a history of myocardial infarction (MI) are at particular risk. Concurrent alterations in myocardial structure & autonomic tone appear important for the development of the arrhythmias leading to SCD.

Given the grave consequences of SCD, an ideal testing procedure should identify most of those at risk (sensitive) & correctly classify risk (accurate). Since >90% of patients who suffer serious arrhythmias post-MI have at least mild left ventricular (LV) dysfunction (ejection fraction [EF] <0.50) this is an optimal group to study.

While noninvasive tests have been developed to estimate SCD risk, prior approaches have failed to: 1) identify the majority of patients at risk for serious arrhythmias (insensitive), 2) evaluate temporal changes in parameters, 3) identify the optimal timing for risk assessment post-MI, & 4) develop a widely-applicable screening tool. This has resulted in a failure to delivery effective therapies (e.g., defibrillator) in a cost-effective manner.

Hypotheses. Primary: Concurrent evaluation of electrical structure & autonomic tone will accurately identify most post-MI patients at risk of serious arrhythmic events. Secondary: 1) assessment later (16 weeks) provides more prognostic information than assessment early post-MI (4 weeks), 2) a single multi-parameter test procedure can be developed, and 3) individually, repolarization alternans provides the most prognostic information.

Methods. 350 persons with a recent MI (<31 days) & EF <0.50 will undergo testing early (4 weeks), intermediate (8 weeks) & late (16 weeks) post-MI.

Four techniques assess cardiac structure (spectral T-wave alternans [TWA], modified moving average TWA; signal-averaged [SA] ECG) & nuclear ejection fraction. Three others evaluate autonomic tone (baroreceptor sensitivity [BRS], heart rate variability [HRV], and Heart Rate Turbulence [HRT]).

Data Collection & Outcomes. Patients will be recruited over 24 months & followed biannually for four years. Committee (blinded) endpoint classification & central laboratory data analysis will be utilized. A composite of resuscitated cardiac arrest and cardiac mortality is the primary outcome. The components (resuscitated / non-resuscitated cardiac arrest and cardiac death) are secondary outcomes.

Statistical Aspects & Sample Size. Standard methods of description & analysis will be used. The capacity to accurately identify most patients at risk for serious arrhythmias will be evaluated using Cox multivariate models. The primary model will include age, sex, EF at 8 wks & important baseline medication use.

Since multivariate modeling requires lower (more sensitive) dichotomy limits the following will be used: spectral TWA positivity will be defined as a non-negative test. SA-ECG QRS width >104 msec will be labeled as abnormal. For HRV, SDNN values <105 msec will be considered abnormal. For BRS, values <6.1 msec per mmHg will indicate impairment. For HRT abnormalities in T-onset & / or T-slope will be considered abnormal. Receiver operating characteristic curves will be used to identify a cut-point for modified moving average TWA.

Assuming a 5 year 20% rate of the composite arrhythmias in patients with positive test results, we have 85% power to detect a 2.5-fold higher risk in patients with abnormalities than those without these abnormalities.

Relevance. This is the first large prospective study to evaluate the utility of concurrent structural & autonomic tone assessment in predicting the development of serious arrhythmias after an MI.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MI <31 days, based upon elevated cardiac-specific CK (total CK-MB mass >7ng/mL or CK-MB/total CK ≥ 2.5%) or troponin-T (> 0.1 ng/ml)144) plus
* clinical symptoms or ECG evidence of myocardial injury (ST deviation ≥ 1 mm in 2, contiguous leads or new/previously undocumented Q waves)144, &
* left ventricular ejection fraction ≤ 0.40 within 48 hrs or ≤ 0.50 beyond 48 hrs of MI using (echocardiography, radionuclide or contrast angiography) &
* Sinus rhythm at the time of enrollment.

Exclusion Criteria:

* Geographic isolation or inability to return for follow-up,
* Comorbid illness likely to cause death within 24 months,
* Inability to complete a submaximal exercise test (e.g., urgent CABG),
* Class I indication for a defibrillator (e.g., VF or sustained VT > 48 hours of index MI), or
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2001-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek V Exner, MD, MPH, Principal Investigator — Libin Cardiovascular Institute of Alberta, University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Result] Exner DV, Kavanagh KM, Slawnych MP, Mitchell LB, Ramadan D, Aggarwal SG, Noullett C, Van Schaik A, Mitchell RT, Shibata MA, Gulamhussein S, McMeekin J, Tymchak W, Schnell G, Gillis AM, Sheldon RS, Fick GH, Duff HJ; REFINE Investigators. Noninvasive risk assessment early after a myocardial infarction the REFINE study. J Am Coll Cardiol. 2007 Dec 11;50(24):2275-84. doi: 10.1016/j.jacc.2007.08.042. Epub 2007 Nov 26. PMID 18068035
- [Derived] Slawnych MP, Nieminen T, Kahonen M, Kavanagh KM, Lehtimaki T, Ramadan D, Viik J, Aggarwal SG, Lehtinen R, Ellis L, Nikus K, Exner DV; REFINE (Risk Estimation Following Infarction Noninvasive Evaluation); FINCAVAS (Finnish Cardiovascular Study) Investigators. Post-exercise assessment of cardiac repolarization alternans in patients with coronary artery disease using the modified moving average method. J Am Coll Cardiol. 2009 Mar 31;53(13):1130-7. doi: 10.1016/j.jacc.2008.12.026. PMID 19324258